CLINICAL TRIAL: NCT06888440
Title: Clinical Effects of Zinc-containing Stents on Gingivitis: a Randomized Controlled Trial
Brief Title: Zinc Stents for the Treatment of Gingivitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Cenk Haytac, Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CukurovaU-dhf12
Record Dates: First submitted 2025-03-14; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Gingivitis; Chronic
Keywords: gingivitis; zinc; treatment
MeSH Terms: conditions — Gingivitis; Bronchiolitis Obliterans Syndrome | interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- zinc containing stent (Experimental): This group will use zinc containing stent after scaling.
  Interventions: Procedure: scaling and zinc stents
- placebo stent (Placebo Comparator): This group will use placebo stent after scaling.
  Interventions: Procedure: scaling and placebo stents

INTERVENTIONS:
Procedure: scaling and zinc stents — this group will receive scaling and zinc containing stents
  Arms: zinc containing stent
Procedure: scaling and placebo stents — this group will receive scaling and placebo stents
  Arms: placebo stent

SUMMARY:
Background This study investigates the effects of zinc-containing stents on gingival inflammation, bleeding, and plaque regrowth in gingivitis patients.

Methods A randomized, double-blind, placebo-controlled study was conducted at Çukurova University, enrolling 42 systemically healthy gingivitis patients aged 18-30. Participants were assigned to either a test group (zinc-containing stents) or a control group (placebo stents) and instructed to wear their stents for at least 12 hours daily for four weeks. Clinical measurements, including Gingival Index (GI), Plaque Index (PI), and Bleeding on Probing (BOP), were assessed at baseline, and at the 2nd, 4th, and 8th weeks. Statistical analysis was performed using IBM SPSS and RStudio.

ELIGIBILITY:
Inclusion Criteria:

* Presence of plaque-induced gingivitis [bleeding on gentle probing at >30% of sites examined and a gingival index (GI) of at least 1 at >60% of sites examined],
* Plaque index (PI) of ≥ 2 according to the modified Quigley&Hein index,
* 18-30 years old,
* At least 20 natural teeth,
* Systemically healthy.

Exclusion Criteria:

* Pocket probing depth (PPD) of ≥4 mm,
* Interdental clinical attachment loss (CAL) detectable at ≥2 nonadjacent teeth or displaying buccal/oral CAL ≥3 mm coupled with PD ≥3 mm
* Subjects with a history of allergies to Zinc,
* The presence of hematologic disorders or any other systemic illness,
* Pregnancy and breastfeeding,
* Current orthodontic treatment,
* History of periodontal therapy,
* Use of antibiotics or anti-inflammatory medication within the preceding 6 months,
* Smoking.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Gingival index | Baseline, 2nd week, 4th week, 8th week
  0- Normal gingiva;
  1. Mild inflammation with slight color change, mild alteration of gingival surface structure and no bleeding on probing;
  2. Moderate inflammation with edema, redness, swelling and bleeding on probing;
  3. Severe inflammation with marked edema and redness, ulceration and tendency to bleed spontaneously.

SECONDARY OUTCOMES:
Plaque index | Baseline, 2nd week, 4th week, 8th week
  0- No plaque;
  1. Separate spots of plaque at the cervical margin of the tooth;
  2. A thin, continuous band of plaque at the cervical margin;
  3. A band of plaque wider than 1 mm but covering less than one-third of the tooth; 4 - plaque covering more than one-third and less than two-thirds of thecrown;
  4. Plaque covering more than two thirds of the crown.
Bleeding on probing | Baseline, 2nd week, 4th week, 8th week
  The bleeding on probing was be measured by using a periodontal probe at six sites per tooth and will be recorded as (+) or (-).

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Cenk Haytac, Professor, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University Faculty of Dentistry, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alkaya B, Kayhan HG, Demirbilek F, Sahin M, Totik N, Ozcan M, Teughels W. Clinical Effects of Zinc-containing Stents on Gingivitis: A Randomised Controlled Trial. Oral Health Prev Dent. 2025 Sep 26;23:577-584. doi: 10.3290/j.ohpd.c_2275. PMID 41001958